CLINICAL TRIAL: NCT02483559
Title: Seeing the World Through Assorted Glasses (SWAG)
Brief Title: Seeing the World Through Assorted Glasses
Acronym: SWAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Eric Youngstrom, PhD, Professor of Psychology and Psychiatry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 15-0389
Record Dates: First submitted 2015-06-13; First posted 2015-06-29 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Sleep
Keywords: Sleep; Photoreceptor Cells, Vertebrate; Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amber Lenses (Other): Participants will be randomized to participate in the amber lens condition first or second. Outcome measures to assess the effects of wearing amber lenses to block the blue light spectrum of light includes mood and sleep rating questionnaires (Positive and Negative Affect Scale, PANAS; Leeds Sleep Evaluation Questionnaire) as well as measuring the levels of melatonin the body is producing while wearing the glasses.
  Interventions: Other: Amber Lenses
- Placebo Lenses (Other): Participants will be randomized to participate in the placebo lens condition first or second. Outcome measures to assess the effects of wearing placebo lenses to allow all spectrums of light includes mood and sleep rating questionnaires (Positive and Negative Affect Scale, PANAS; Leeds Sleep Evaluation Questionnaire) as well as measuring the levels of melatonin the body is producing while wearing the glasses.
  Interventions: Other: Placebo Lenses

INTERVENTIONS:
Other: Amber Lenses — Glasses fitted with amber lenses that block the blue spectrum of light (~470 nm) to be worn prior to desired sleep onset time.
  Arms: Amber Lenses
Other: Placebo Lenses — Glasses fitted with placebo lenses that allow all visible spectrum of light to be worn prior to desired sleep onset time.
  Arms: Placebo Lenses

SUMMARY:
The purpose of the study is to test the use of amber glasses at night as a method to block blue light from the eye, allowing the brain to produce a dim-light melatonin onset. The investigators hypothesize that blue-blocking will produce measurable benefits in subjectively and objectively rated sleep quality and mood as well as salivary melatonin levels during the night.

DETAILED DESCRIPTION:
Participants will complete a self-report battery containing measures of sleep quality, morningness-eveningness chronotype, and mood. Participants will then wear a wrist-worn accelerometer for 14 days to objectively record activity level and sleep quality. Participants will also fill out a daily sleep log and short self-report measures assessing sleep and mood. On days 4-7 and 11-14 of the study the participants will wear either amber or placebo control lenses prior to sleep onset in a randomized crossover design (i.e., participants will be randomized to wear either amber lenses or placebo lenses for the first part of the protocol and then switch to wear the opposite lenses for the second part of the protocol). Participants will spend nights 7 and 14 of the study in a sleep laboratory in order to obtain hourly melatonin samples and wear a wrist sleep monitor to non-invasively and objectively measure sleep state and quality using peripheral arterial tone and oxygen perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Good physical health
* Proficiency in written and spoken English
* Reported average total sleep time <9 hours (so nights spent in sleep lab will not result in sleep deprivation)

Exclusion Criteria:

* Taking regular medication affecting sleep and/or mood
* Travel across more than two time zones within the past month
* Smoke > 5 cigarettes per day
* Excessive caffeine use (>2 cups at one time or >500 mg daily)
* No current Axis I Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Disorder
* No current use of street drugs
* No history of sleep disorder/bipolar disorder/psychosis/seizure disorder/chronic medical condition
* Night shift work within the past 2 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Increase dim-light melatonin production | 4 days
  Hourly saliva samples will be collected from participants at the end of each 4 night interval in order to measure levels of melatonin production.

SECONDARY OUTCOMES:
Improved subjective self-reported mood | 4 days
  Participants will complete the Positive and Negative Affect Scale (PANAS) on a daily basis to measure self-reported mood.
Improved objective measures of sleep | 4 days
  Participants will complete nights in the sleep lab while wearing a watch device to measure arterial tone in order to objectively measure time spent in different sleep stages.
Improved subjective self-reported sleep quality | 4 days
  Participants will complete the Leeds Sleep Evaluation in order to assess self-report of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Youngstrom, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States